CLINICAL TRIAL: NCT06028243
Title: Assessment of the Effectiveness of the Healthy Living Awareness Program for the Prevention of Osteoporosis Based on the Information- Motivation- Behavioral Skills Model in University Students: A Randomized Controlled Trial
Brief Title: Awareness Model in Prevention of Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Sibel Peksoy Kaya, Asst. Prof., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-12
Record Dates: First submitted 2023-08-17; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Osteoporosis; University Students; Healthy Lifestyle
Keywords: Osteoporosis; Health Behaviors; Health Beliefs; Motivation; Physical Activity; Program Planning; Self-Efficacy; Health Information
MeSH Terms: conditions — Osteoporosis; Health Behavior; Motor Activity

STUDY DESIGN:
Masking Description: Blinding in the study was not feasible. Blinding could not be performed because the researchers were aware of the interventions and carried out the implementation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB) was implemented in three stages.
  Information stage: The researchers provided the intervention group participants with online training in healthy living awareness to prevent osteoporosis. The training consisted of four sections: osteoporosis and diagnosis-treatment methods, current approaches to the prevention of osteoporosis, osteoporosis and nutrition, and osteoporosis and physical exercise. At the end of the training, the participants were informed about the healthy life diary and record.
  Motivation stage: The researchers regularly texted reminder notifications concerning the prevention of osteoporosis. The records in their diaries were reviewed. The researchers provided individual counseling to the participants by telephone.
  Behavior skills stage: The target behavior skills were improved self-efficacy in doing weight-bearing exercises, taking calcium, and engaging in physical activity.
  Interventions: Other: The Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB)- Information stage; Other: The Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB)- Motivation stage; Behavioral: The Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB)- Behavior skills stage
- Control Group (No Intervention): The control group was not trained. Data collection forms applied to the intervention group were also applied to the control group simultaneously.

INTERVENTIONS:
Other: The Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB)- Information stage — The researchers provided the intervention group participants with online training in healthy living awareness to prevent osteoporosis (400 minutes and two days). They held the training at all participants' convenience outside the class hours. The training consisted of four sections: (1) osteoporosis and diagnosis-treatment methods, (2) current approaches to the prevention of osteoporosis, (3) osteoporosis and nutrition, and (4) osteoporosis and physical exercise. The researchers employed interactive teaching methods and consulted three experts to prepare PowerPoint presentations. At the end of the training, the researchers taught the intervention group participants how to fill out the healthy life diary, such as calculating daily calcium intake. The researchers texted the intervention group participants all training videos on WhatsApp to allow them to watch them again.
  Arms: Intervention Group
Other: The Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB)- Motivation stage — The researchers regularly texted (WhatsApp) spot and reminder notifications concerning the prevention of osteoporosis. They asked them to assess the health behaviors they recorded in their diaries every week (daily calcium intake, weekly exercise duration, etc.) and the problems they experienced during the process. The researchers provided individual counseling to the participants by telephone (combating smoking, exercise barriers, food exchange for calcium sources, etc.)
  Arms: Intervention Group
Behavioral: The Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB)- Behavior skills stage — The target behavior skills were improved self-efficacy in doing weight-bearing exercises, taking calcium, and engaging in physical activity.
  Arms: Intervention Group

SUMMARY:
This study investigated the effectiveness of a Healthy Living Awareness Program for the Prevention of Osteoporosis based on the Information-Motivation-Behavioral Skills Model (HLAPPO-IMB) in university students. The study adopted a randomized controlled trial intervention pretest, posttest, and follow-up research design. Participants were randomized into intervention (n=43) and control groups (n=44). Data were collected using a personal information form, the Osteoporosis Knowledge Test, the Osteoporosis Health Belief Scale, the Osteoporosis Self-Effective Scale, and the International Physical Activity Questionnaire Short Form.

The primary outcome measure was the participants' knowledge and health beliefs about osteoporosis. The secondary outcome measure was the participants' healthy lifestyle behavior skills (self-efficacy in weight-bearing exercises, taking calcium, and engaging in physical activity).

Research questions (RQ) RQ1: Does "Healthy Living Awareness Program for the Prevention of Osteoporosis based on the Information-Motivation-Behavioral Skills Model" expand participants' knowledge of osteoporosis? RQ2: Does "Healthy Living Awareness Program for the Prevention of Osteoporosis based on the Information-Motivation-Behavioral Skills Model" enhance participants' health beliefs? RQ3: Does "Healthy Living Awareness Program for the Prevention of Osteoporosis based on the Information-Motivation-Behavioral Skills Model" improve participants' self-efficacy in doing weight-bearing exercises and taking calcium? RQ4: Does "Healthy Living Awareness Program for the Prevention of Osteoporosis based on the Information-Motivation-Behavioral Skills Model" improve participants' self-efficacy in engaging in physical activity?

DETAILED DESCRIPTION:
This study adopted a randomized controlled trial pretest, posttest, and follow-up research design. The study was conducted between March and August 2021 at a public university in Türkiye. The study adhered to the CONSORT (Consolidated Standards of Reporting Trials) guidelines. Participants were randomized into intervention and control groups. Eligible students were randomized to intervention group or control group using block randomization technique. Blinding in the study was not feasible. Blinding could not be performed because the researchers were aware of the interventions and carried out the implementation. The intervention group attended the HLAPPO-IMB, which had three stages: information, motivation, and behavioral skills development. The control group did not undergo the intervention.

The study population consisted of 125 fifth-semester nursing students in the fall term of the 2020-2021 academic year. The undergraduate nursing programs in Türkiye are eight-semester programs. The mean Osteoporosis Knowledge Test (OKT) scores were used to determine the sample size. Power analyses were performed based on the difference between two independent means by G*Power 3.1.9.7. A power analysis was performed to determine the sample size in line with the literature [OKT: experimental group X̅±SD: 18.95±4.98 and control group X̅±SD: 15.18±3.88]. The results showed that a sample of 76 would be large enough to detect significant differences (0.84 effect size, 0.05 level of error, and 95% power). All students who met the inclusion criteria were recruited to avoid missing data. The first sample consisted of 87 participants, who were randomized to intervention (n=43) and control (n=44) groups. However, one student from the intervention group declined to participate. Therefore, the final sample consisted of 86 participants.

The data were collected using a personal information form, the Osteoporosis Knowledge Test (OKT), the Osteoporosis Health Belief Scale (OHSB), the Osteoporosis Self-Effective Scale (OSES), and the International Physical Activity Questionnaire Short Form (IPAQ-SF).

The personal information form: This form was prepared by the researchers. The form consisted of 30 items on sociodemographic characteristics and factors that might affect bone mineral density. Each participant's BMI, body weight, and body height were calculated based on his/her self-report.

Osteoporosis knowledge test: The instrument consists of 24 items. The total score ranges from 0 to 24, with higher scores indicating more osteoporosis-related knowledge.

Osteoporosis health belief scale: The instrument consists of 42 items rated on a Likert-type scale. The total score ranges from 42 to 210, with higher scores indicating more positive health beliefs about osteoporosis.

Osteoporosis self-effective scale: The scale consists of 12 items and two subscales: The Osteoporosis Self-Efficacy Exercise Scale (six items: starting an exercise program, changing exercise habits, doing appropriate exercise, etc.) and the Osteoporosis Self-Efficacy Calcium Scale (six items: increasing calcium intake, choosing calcium-rich foods, maintaining dietary calcium intake, etc.). The total score of each subscale ranges from 0 to 600. The total score ranges from 0 to 1200, with higher scores indicating better self-efficacy in weight-bearing exercises and taking calcium.

International physical activity questionnaire short form: The form consists of seven items on physical activity. The total score is the "Metabolic Equivalent of Task minute/week (MET min/week)." The total score is calculated as "MET min/week" by multiplying the minute, day, and MET values. Physical activity levels are classified as low (<600 MET min/week), moderate (600-3000 MET min/week), or high (>3000 MET min/week) according to the total MET min/week values.

Healthy life diary: The researchers developed the Healthy Life Diary to monitor the intervention group participants' healthy lifestyle behaviors to protect themselves from osteoporosis. The intervention group participants filled out the diary regularly and noted their daily calcium intake, type and duration of exercise, duration and time of sunlight exposure, and amount of tobacco, coffee, tea, cola, etc.

Procedure: The data were collected online because of the COVID-19 pandemic. The researchers briefed students on the research procedure and texted them a link to the survey on WhatsApp. The first page of the survey was a consent form. After obtaining informed consent, the researchers directed all students who agreed to participate to the inclusion criteria section. Students are a vulnerable population. Thus, the researchers took measures to ensure students would not feel coerced to participate. The researchers informed all students about the research purpose and procedure. Participation was voluntary. The researchers kept all personal information confidential. All participants had pseudonyms.

Healthy living awareness program for the prevention of osteoporosis: The intervention group participants underwent the Healthy Living Awareness Program for the Prevention of Osteoporosis (HLAPPO-IMB) in three stages based on IMB.

Information stage: The researchers provided the intervention group participants with online training in healthy living awareness to prevent osteoporosis (400 minutes and two days). They held the training at all participants' convenience outside the class hours. The training consisted of four sections: osteoporosis and diagnosis-treatment methods, current approaches to the prevention of osteoporosis, osteoporosis and nutrition, and osteoporosis and physical exercise. The researchers employed interactive teaching methods and consulted three experts to prepare PowerPoint presentations. At the end of the training, the researchers taught the intervention group participants how to fill out the healthy life diary, such as calculating daily calcium intake. The researchers texted the intervention group participants all training videos on WhatsApp to allow them to watch them again. All participants filled out the OKT and OHSB (posttest) two and three weeks after the training. They filled them out again two months after the posttest (follow-up).

Motivation stage: The researchers regularly texted (WhatsApp) spot and reminder notifications concerning the prevention of osteoporosis. They asked them to assess the health behaviors they recorded in their diaries every week (daily calcium intake, weekly exercise duration, etc.) and the problems they experienced during the process. The researchers provided individual counseling to the participants by telephone (combating smoking, exercise barriers, food exchange for calcium sources, etc.)

Behavior skills stage: The target behavior skills were improved self-efficacy in doing weight-bearing exercises, taking calcium, and engaging in physical activity. The OSES was used to assess participants' self-efficacy to initiate and maintain behavior related to exercise and calcium taking, while the IPAQ-SF was used to assess their physical activity levels.

Data analysis: The data were analyzed using the Statistical Package for Social Sciences. Percentage, mean, and standard deviation were used for descriptive analysis. The categorical variables were analyzed using the Pearson, Fisher χ2, and Marginal Homogeneity tests. The Mann-Whitney U test was used to compare two independent groups. The Wilcoxon Signed Rank test or Friedman nonparametric test was used for dependent measurement comparisons. The effect size (r or Kendall W) was calculated for each comparison. The following limit values were accepted for the interpretation of the effect sizes: r < 0.29 "small effect," r=0.30-0.49 "medium effect," r ≥ 0.50 "large effect." W effect size: <0.39 "small effect," 0.40-0.59 "medium effect,"≥ 0.60 "large effect". The Mann-Whitney U Test was used to compare the difference in age, menarche age, BMI, and scale scores between the groups. The Wilcoxon Signed Rank test was used to compare the pretest and posttest scores. Friedman test was used for repeated measures for dependent groups. Dunn's Bonferroni correction was used to determine the source of the difference.

ELIGIBILITY:
Inclusion Criteria:

* having received no training on osteoporosis before
* having no disability that prevents physical activity

Exclusion Criteria:

* involuntary

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
The effect of the program on the primary outcome-1 (Osteoporosis Knowledge Test) | Pretest: 3 weeks, Completion of training: 2 weeks, Posttest: 2 weeks (2-3 weeks after training), Follow-up: 2 weeks (2 months after posttest). Total period of research: 20 weeks. Total application time of this scale: 7weeks.
  Osteoporosis Knowledge Test consists of 24 items. The total score ranges from 0 to 24, with higher scores indicating more osteoporosis-related knowledge.
  Osteoporosis Knowledge Test with Osteoporosis Health Belief Scale was applied three times (pretest, posttest and follow-up) to the intervention and control groups. Training was given to the intervention group after completing the Osteoporosis Knowledge Test (with other scales) as a pretest. After the training, it was applied to the participants as a posttest and follow-up. All participants filled out the Osteoporosis Knowledge Test with Osteoporosis Health Belief Scale (posttest) two and three weeks after the training. They filled them out again two months after the posttest (follow-up).
  In the study protocol, pretest postest and follow up times are given in detail.
The effect of the program on the primary outcome-2 (Osteoporosis Health Belief Scale) | Pretest: 3 weeks, Completion of training: 2 weeks, Posttest: 2 weeks (2-3 weeks after training), Follow-up: 2 weeks (2 months after posttest). Total period of research: 20 weeks. Total application time of this scale: 7weeks.
  Osteoporosis Health Belief Scale consists of 42 items rated on a Likert-type scale. The total score ranges from 42 to 210, with higher scores indicating more positive health beliefs about osteoporosis.
  Osteoporosis Health Belief Scale with Osteoporosis Knowledge Test was applied three times (pretest, posttest and follow-up) to the intervention and control groups. Training was given to the intervention group after completing the Osteoporosis Health Belief Scale (with other scales) as a pretest. After the training, it was applied to the participants as a posttest and follow-up. All participants filled out the Osteoporosis Health Belief Scale with Osteoporosis Knowledge Test (posttest) two and three weeks after the training. They filled them out again two months after the posttest (follow-up).

SECONDARY OUTCOMES:
The effect of the program on the secondary outcome-1 (Osteoporosis Self-Effective Scale) | Pretest: 3 weeks, training and follow-up period: 15 weeks, Follow-up: 2 weeks. Total period of research: 20 weeks. Total application time of this scale: 5 weeks.
  Osteoporosis Self-Effective Scale consists of 12 items and two subscales: The Osteoporosis Self-Efficacy Exercise Scale (six items: starting an exercise program, changing exercise habits, doing appropriate exercise, etc.) and the Osteoporosis Self-Efficacy Calcium Scale (six items: increasing calcium intake, choosing calcium-rich foods, maintaining dietary calcium intake, etc.). The total score of each subscale ranges from 0 to 600. The total score ranges from 0 to 1200, with higher scores indicating better self-efficacy in weight-bearing exercises and taking calcium.
  Osteoporosis Self-Effective Scale was applied twice (pretest and follow-up) with International Physical Activity Questionnaire Short Form to the study groups. It was applied as a pretest with other scales. It was applied as a follow-up 13 weeks after the training.
The effect of the program on the primary outcome-2 (International Physical Activity Questionnaire Short Form) | Pretest: 3 weeks, training and follow-up period: 15 weeks, Follow-up: 2 weeks. Total period of research: 20 weeks. Total application time of this scale: 5 weeks.
  International Physical Activity Questionnaire Short Form consists of seven items on physical activity. The total score is the "Metabolic Equivalent of Task minute/week)." The total score is calculated as "Metabolic Equivalent of Task minute/week " by multiplying the minute, day, and Metabolic Equivalent of Task values. Physical activity levels are classified as low, moderate, or high according to the total Metabolic Equivalent of Task min/week values. International Physical Activity Questionnaire Short Form was applied twice (pretest and follow-up) with Osteoporosis Self-Effective Scale to the study groups. It was applied as a pretest with other scales. It was applied as a follow-up 13 weeks after the training.

CONTACTS AND LOCATIONS:
Overall Officials: SİBEL PEKSOY KAYA, Asst. Prof., Principal Investigator — ANKARA YILDIRIM BEYAZIT UNIVERSITY, ANKARA, TURKEY; SENA KAPLAN, Prof. Dr., Study Director — ANKARA YILDIRIM BEYAZIT UNIVERSITY, ANKARA, TURKEY; ESRA BAŞKAYA, Dr., Study Director — ANKARA YILDIRIM BEYAZIT UNIVERSITY, ANKARA, TURKEY
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Background] Aktas O, Kaplan S, Sezer N. An assessment of the relation between bone mineral density and clinic-demographic properties and life quality during postmenopausal period. J Back Musculoskelet Rehabil. 2018;31(5):803-810. doi: 10.3233/BMR-170933. PMID 29865030
- [Background] Alpar, R. (2022). Spor Sağlık ve Eğitim Bilimlerinden Örneklerle Uygulamalı İstatistik ve Geçerlik Güvenirlik; (7th edition). Ankara: Detay Yayıncılık.
- [Background] Bahrami Z, Zarani F. Application of the Information-Motivation and Behavioral Skills (IMB) model in risky sexual behaviors amongst male students. J Infect Public Health. 2015 Mar-Apr;8(2):207-13. doi: 10.1016/j.jiph.2014.09.005. Epub 2014 Nov 22. PMID 25466597
- [Background] Barley E, Lawson V. Using health psychology to help patients: theories of behaviour change. Br J Nurs. 2016 Sep 8;25(16):924-7. doi: 10.12968/bjon.2016.25.16.924. PMID 27615529
- [Background] Bonjour JP, Theintz G, Law F, Slosman D, Rizzoli R. Peak bone mass. Osteoporos Int. 1994;4 Suppl 1:7-13. doi: 10.1007/BF01623429. PMID 8081064
- [Background] Bonjour, P., Compston, J., Dawson-Hughes, B., Delmas, P., Lyon, H. E. H., Ms, F., Johansson, H., Kanis, J. A., Lau, E., Yuen, L., Centre, H., Kong, H., Dr, C., Lindsay, R., Mcclung, M. R., Oden, A., Pfleger, B., Teilen, M. G., Clark Hospital De Especialidades, P., … Toroptsova, N. (2007). Assessment of Osteoporosis at The Primary Health Care Level. www.who.int/chp/topics/rheumatic/en/index.html
- [Background] Cooper, C., & Ferrari, S. (2019). IOF Compendium of Osteoporosis (2nd Edition). Switzerland: International Osteoporosis Foundation.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] EQUATOR guidelines. (2020). Checklist for reporting a randomised trial. Retrieved from: https://www.goodreports.org/reporting-checklists/consort/
- [Background] Haleem A, Javaid M, Vaishya R. Effects of COVID-19 pandemic in daily life. Curr Med Res Pract. 2020 Mar-Apr;10(2):78-79. doi: 10.1016/j.cmrp.2020.03.011. Epub 2020 Apr 3. No abstract available. PMID 32292804
- [Background] Hernlund E, Svedbom A, Ivergard M, Compston J, Cooper C, Stenmark J, McCloskey EV, Jonsson B, Kanis JA. Osteoporosis in the European Union: medical management, epidemiology and economic burden. A report prepared in collaboration with the International Osteoporosis Foundation (IOF) and the European Federation of Pharmaceutical Industry Associations (EFPIA). Arch Osteoporos. 2013;8(1):136. doi: 10.1007/s11657-013-0136-1. Epub 2013 Oct 11. PMID 24113837
- [Background] Hosseini, Z., Karimi, Z., Mohebi, S., Reza Sharifirad, G., Rahbar, A., & Gharlipour, Z. (2017). Nutritional preventive behavior of osteoporosis in female students: Applying health belief model (HBM). International Journal of Pediatrics, 5(37). https://doi.org/10.22038/ijp.2016.7560
- [Background] Kılıç, D., & Erci, B. (2010). The reliability and validity of the osteoporosis health belief scale, osteoporosis self-efficacy scale and osteoporosis knowledge test. Journal of Anatolia Nursing and Health Sciences, 7(2), 89-102. https://dergipark.org.tr/en/pub/ataunihem/issue/2627/33798
- [Background] Kim, K., Horan, M., & Gendler, P. (1991). Osteoporosis Knowledge Test, Osteoporosis Health Belief Scale, and Osteoporosis Self-efficacy Scale Allendale: MI: Grand Valley State University; Allendale. Masterson R. A descript.
- [Background] Kline J, Tang A, Levin B. Smoking, alcohol and caffeine in relation to two hormonal indicators of ovarian age during the reproductive years. Maturitas. 2016 Oct;92:115-122. doi: 10.1016/j.maturitas.2016.07.010. Epub 2016 Jul 21. PMID 27621248
- [Background] Majumdar SR, Lier DA, McAlister FA, Johnson JA, Rowe BH, Beaupre LA. Cost-Effectiveness of Osteoporosis Interventions to Improve Quality of Care After Upper Extremity Fracture: Results From a Randomized Trial (C-STOP Trial). J Bone Miner Res. 2019 Jul;34(7):1220-1228. doi: 10.1002/jbmr.3699. Epub 2019 Mar 18. PMID 30779861
- [Background] Oka R, Ohira M, Suzuki S, Yoshida T, Koide H, Tanaka T, Tatsuno I. Fracture risk assessment tool (FRAX) and for the diagnosis of osteoporosis in Japanese middle-aged and elderly women: Chiba bone survey. Endocr J. 2018 Feb 26;65(2):193-202. doi: 10.1507/endocrj.EJ17-0331. Epub 2017 Nov 18. PMID 29151451
- [Background] Pouresmaeili F, Kamalidehghan B, Kamarehei M, Goh YM. A comprehensive overview on osteoporosis and its risk factors. Ther Clin Risk Manag. 2018 Nov 6;14:2029-2049. doi: 10.2147/TCRM.S138000. eCollection 2018. PMID 30464484
- [Background] Qi BB, Resnick B, Smeltzer SC, Bausell B. Self-efficacy program to prevent osteoporosis among Chinese immigrants: a randomized controlled trial. Nurs Res. 2011 Nov-Dec;60(6):393-404. doi: 10.1097/NNR.0b013e3182337dc3. PMID 22048557
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] TC. Sağlık Bakanlığı Halk Sağlığı Kurumu. (2016). Türkiye Beslenme Rehberi 2015 (TÜBER). T.C. Sağlık Bakanlığı Yayın No: 1031. Ankara.
- [Background] Ficek K, Rajca J, Cholewinski J, Racut A, Gwiazdon P, Przednowek K, Hajduk G. Analysis of intercondylar notch size and shape in patients with cyclops syndrome after anterior cruciate ligament reconstruction. J Orthop Surg Res. 2021 Sep 8;16(1):554. doi: 10.1186/s13018-021-02706-w. PMID 34496898
- [Background] Si M, Su X, Jiang Y, Wang W, Zhang X, Gu X, Ma L, Li J, Zhang S, Ren Z, Liu Y, Qiao Y. Effect of an IMB Model-Based Education on the Acceptability of HPV Vaccination Among College Girls in Mainland China: A Cluster RCT. Cancer Control. 2022 Jan-Dec;29:10732748211070719. doi: 10.1177/10732748211070719. PMID 35088609
- [Background] Tsamlag L, Wang H, Shen Q, Shi Y, Zhang S, Chang R, Liu X, Shen T, Cai Y. Applying the information-motivation-behavioral model to explore the influencing factors of self-management behavior among osteoporosis patients. BMC Public Health. 2020 Feb 6;20(1):198. doi: 10.1186/s12889-020-8292-x. PMID 32028930
- [Background] Tuzun S, Eskiyurt N, Akarirmak U, Saridogan M, Senocak M, Johansson H, Kanis JA; Turkish Osteoporosis Society. Incidence of hip fracture and prevalence of osteoporosis in Turkey: the FRACTURK study. Osteoporos Int. 2012 Mar;23(3):949-55. doi: 10.1007/s00198-011-1655-5. Epub 2011 May 19. PMID 21594756
- [Background] Upadhyaya GK, Iyengar K, Jain VK, Vaishya R. Challenges and strategies in management of osteoporosis and fragility fracture care during COVID-19 pandemic. J Orthop. 2020 Jun 2;21:287-290. doi: 10.1016/j.jor.2020.06.001. eCollection 2020 Sep-Oct. PMID 32523258
- [Background] World Health Organization (WHO). A healthy lifestyle-WHO recommendations (2023). Retrieved from: https://www.who.int/europe/news-room/fact-sheets/item/a-healthy-lifestyle---who-recommendations
- [Background] Yekefallah, L., Dehghankar, L., Aliakbari, M., & Mafi, M. (2019). Lifestyle and preventive behaviors of osteoporosis among women of reproductive age in Qazvin-Iran: A cross sectional study. Social Health and Behavior, 2(2), 70. https://doi.org/10.4103/SHB.SHB_50_18
- [Result] Abay H, Kaplan S. Evaluation of the effectiveness of a training program for coping with PMS symptoms based on IMB model in university students. Women Health. 2021 Jul;61(6):550-561. doi: 10.1080/03630242.2021.1927286. Epub 2021 Jun 1. PMID 34074223
- [Result] Fisher JD, Fisher WA. Changing AIDS-risk behavior. Psychol Bull. 1992 May;111(3):455-74. doi: 10.1037/0033-2909.111.3.455. PMID 1594721
- [Result] Hong SY, Jun SY. Community Capacity Building Exercise Maintenance Program for Frail Elderly Women. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Sep;11(3):166-173. doi: 10.1016/j.anr.2017.06.001. Epub 2017 Aug 10. PMID 28991596
- [Result] Kim, Y. il, & Park, J. S. (2017). Development and evaluation of a joint health self-management program for the elderly with knee osteoarthritis in communities: applying the IMB model. Research in Community and Public Health Nursing, 28(1), 55-68. https://doi.org/10.12799/JKACHN.2017.28.1.55
- [Result] Lee Y, Kim DH. A preliminary study on the effects of an osteoporosis prevention program based on an Information-Motivation-Behavioral skill model in older adult women: A cluster randomized controlled trial. Geriatr Nurs. 2022 May-Jun;45:55-63. doi: 10.1016/j.gerinurse.2022.03.001. Epub 2022 Mar 22. PMID 35334422
- [Result] Morton, M., & Montgomery, P. (2011). Youth empowerment programs for improving self-efficacy and self-esteem of adolescents. Campbell Systematic Reviews, 7(1), 1-80. https://doi.org/10.4073/CSR.2011.5
- [Result] Panahi R, Siboni FS, Kheiri M, Ghoozlu KJ, Shafaei M, Dehghankar L. Promoting the adoption of behaviors to prevent osteoporosis using the health belief model integrated with health literacy: quasi-experimental intervention study. BMC Public Health. 2021 Dec 7;21(1):2221. doi: 10.1186/s12889-021-12300-8. PMID 34872550
- [Result] Park SJ, Jung JH, Kim MS, Lee HJ. High dairy products intake reduces osteoporosis risk in Korean postmenopausal women: A 4 year follow-up study. Nutr Res Pract. 2018 Oct;12(5):436-442. doi: 10.4162/nrp.2018.12.5.436. Epub 2018 Oct 1. PMID 30323911
- [Result] Shawashi, T. O., & Darawad, M. (2020). Osteoporosis knowledge, beliefs and self-efficacy among female university students: a descriptive study. The Open Nursing Journal, 14(1), 211-219. https://doi.org/10.2174/1874434602014010211
- [Result] Shell DF, Newman IM, Perry CM, Folsom AR. Changing intentions to use smokeless tobacco: an application of the IMB model. Am J Health Behav. 2011 Sep;35(5):568-80. doi: 10.5993/ajhb.35.5.6. PMID 22040618
- [Result] Tastekin Ouyaba A, Ozyurek P, Sevil U. The effect of an information, motivation, and behavioral skills model intervention on young women's intention to get an HPV vaccine. Psychol Health Med. 2023 Mar;28(3):732-742. doi: 10.1080/13548506.2021.1975780. Epub 2021 Sep 5. PMID 34486461
- [Result] Yeager DS, Dahl RE, Dweck CS. Why Interventions to Influence Adolescent Behavior Often Fail but Could Succeed. Perspect Psychol Sci. 2018 Jan;13(1):101-122. doi: 10.1177/1745691617722620. Epub 2017 Dec 12. PMID 29232535
- [Derived] Peksoy-Kaya S, Kaplan S, Baskaya E. A survey of the effect of an information-motivation-behavioral model-based intervention on university students' osteoporosis knowledge, health beliefs, and self-efficacy. Women Health. 2024 Nov-Dec;64(10):870-883. doi: 10.1080/03630242.2024.2422884. Epub 2024 Nov 4. PMID 39496478

DOCUMENTS (1):
  • Study Protocol (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT06028243/Prot_000.pdf